CLINICAL TRIAL: NCT06629116
Title: Study on the Role of Human Serum Albumin in Large Acute Ischemic Stroke of Anterior Circulation After Thrombectomy: A Prospective, Multicenter, Open-label, Endpoint-blinded, Randomized Controlled Trial
Brief Title: Study on the Role of Human Serum Albumin in Large Acute Ischemic Stroke of Anterior Circulation After Thrombectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tingyu-Yi (Other)
Responsible Party: Sponsor-Investigator, Tingyu-Yi, Doctor, Zhangzhou Municipal Hospital
Organization: Zhangzhou Municipal Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Human Serum Albumin
Record Dates: First submitted 2023-10-05; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Ischemia
MeSH Terms: conditions — Brain Ischemia | interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Albumin group (Experimental): Patients with AIS receive intravascular therapy, and within 10 minutes after the surgery, they are administered 100ml of 20% human albumin intravenously (infused within 30 minutes).
  Interventions: Drug: Patients with AIS receive intravascular therapy, and within 10 minutes after the surgery, they are administered 100ml of 20% human albumin intravenously (infused within 30 minutes).
- Control group (No Intervention): Follow the current guidelines for standard conventional treatment.

INTERVENTIONS:
Drug: Patients with AIS receive intravascular therapy, and within 10 minutes after the surgery, they are administered 100ml of 20% human albumin intravenously (infused within 30 minutes). — Whether to administer albumin to AIS patients after intravascular thrombectomy and reperfusion.
  Other Names: Albumin
  Arms: Albumin group

SUMMARY:
This project intends to explore the therapeutic efficacy of human serum albumin in mitigating postoperative cerebral edema and enhancing clinical outcomes following mechanical thrombectomy in patients with acute anterior circulation large-core ischemic stroke.

DETAILED DESCRIPTION:
Human serum albumin is an important biological molecule that plays a critical role in maintaining intracellular osmotic pressure, combating oxidative stress, and suppressing inflammatory responses. Studies have indicated that serum albumin levels gradually decrease in acute-phase stroke patients, accompanied by increased blood-brain barrier disruption. Low albumin levels may exacerbate the progression of cerebral infarction. Furthermore, another study found a correlation between serum albumin levels and the prognosis of AIS. Research has confirmed that human serum albumin may have potential benefits in neuroprotection through mechanisms such as improving microcirculation, reducing oxidative stress, and inhibiting inflammatory responses.

In an experimental animal study of ischemic stroke, researchers discovered that in the middle cerebral artery occlusion (MCAO) model, rats treated with albumin showed significantly reduced neurological function scores and infarct volume compared to the saline group. The mechanism behind this effect may be related to albumin's ability to improve ischemic penumbral blood flow and enhance perfusion in occluded vessels' distal regions. Multiple preclinical studies have suggested that using albumin therapy after vascular recanalization can significantly reduce infarct volume, alleviate brain edema, and improve neurological function, highlighting the neuroprotective role of serum albumin. However, the clinical efficacy of serum albumin in ischemic stroke remains a subject of controversy.

The aim of this study is to investigate the role of human serum albumin in acute anterior circulation large core ischemic stroke after thrombectomy reperfusion, with the hope of providing new insights and methods for clinical treatment. This study will employ a prospective, multicenter, open-label, endpoint-blinded, randomized controlled research design to systematically evaluate the therapeutic effects of human serum albumin in acute anterior circulation large core ischemic stroke after thrombectomy reperfusion. Through clinical observation, imaging assessment, neurofunctional evaluation, and other methods, the investigators will delve into the intervention of human serum albumin in reperfusion injury and its mechanisms in neuroprotection. This research is expected to offer new perspectives and methods for the treatment of patients with acute anterior circulation large core ischemic stroke, provide scientific evidence for clinical practice, and contribute positively to improving patient outcomes and reducing the societal burden.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old.
2. Acute ischemic stroke patients with NIHSS score ≥ 6.
3. Pre-stroke mRS (modified Rankin Scale) score ≤ 1.
4. Onset of symptoms to presentation within 24 hours, including wake-up strokes or strokes without witnessed onset; the time of symptom onset is defined as the "last seen normal" time.
5. Confirmed by CTA/MRA/DSA to have anterior circulation large vessel occlusive ischemic stroke (occlusion of the internal carotid artery or M1 or M2 segments of the middle cerebral artery), responsible for acute ischemic stroke signs and symptoms.
6. ASPECTS (Alberta Stroke Program Early CT Score) on NCCT (non-contrast CT) 3-6 or cerebral perfusion imaging: core infarct volume (rCBF ≤ 30%) 50-100 ml.
7. Achieving vessel reperfusion of mTICI (modified Thrombolysis in Cerebral Infarction) grade 2b or 3 through mechanical thrombectomy.
8. Written informed consent signed by the patient or their legally authorized representative.

Exclusion Criteria:

1. Intracranial hemorrhage confirmed by head CT or MRI.
2. Pre-stroke mRS score > 2.
3. Severe allergy or absolute contraindication to iodine-based contrast agents.
4. Systolic blood pressure > 185 mmHg or diastolic blood pressure > 110 mmHg, and inability to control with antihypertensive medication.
5. Blood glucose < 50 mg/dl (2.8 mmol/L) or > 400 mg/dl (22.2 mmol/L) and difficult to correct.
6. Genetic or acquired bleeding diathesis, deficiency of coagulation factors, or oral anticoagulation with INR > 1.7.
7. Severe renal dysfunction defined as serum creatinine > 3.0 mg/dl (or 265.2 μmol/l) or glomerular filtration rate (GFR) < 30 ml/min, or need for hemodialysis or peritoneal dialysis.
8. Expected life expectancy < 6 months.
9. Anticipated inability of the patient to complete the 90-day follow-up.
10. Suspected aortic dissection.
11. Brain tumors, intracranial aneurysms, or arteriovenous malformations with mass effect on imaging.
12. Neurological or psychiatric disorders affecting the assessment of the disease before the patient's stroke.
13. Pregnancy or reproductive-age women with positive urinary or serum β-human chorionic gonadotropin (HCG) test.
14. Currently participating in other clinical trials that may interfere with the results of this trial.
15. History of allergy to albumin.
16. Need for intermittent or long-term concomitant acute or chronic pulmonary diseases.
17. Congestive heart failure for any reason in the past 6 months or any condition requiring medication, hospitalization, etc., related to heart failure.
18. Symptomatic or diagnosed acute myocardial infarction, or occurrence of acute myocardial infarction within the past 6 months.
19. Other situations that the investigator believes are not suitable for participation or may pose significant risks to the patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Functional independence Rate | From enrollment to the end of treatment at 3 months
  mRS score of 0-2

SECONDARY OUTCOMES:
Rate of independent ambulation | From enrollment to the end of treatment at 3 months
  modified Rankin Scale score of 0-3 scores

OTHER OUTCOMES:
sICH occurrence | within 72 hours after enrollment
  New occurs Intracranial hemorrhage with NIHSS increase >=4 points

CONTACTS AND LOCATIONS:
Overall Officials: Tingyu Yi, Postgraduate, Principal Investigator — zhangzhou Affiliated Hospital to Fujian Medical University , Fujian ,China
Locations (1):
- Zhangzhou Municipal Hospital, Zhangzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
not sure